CLINICAL TRIAL: NCT01206647
Title: Investigation of a Switch From Insulin Therapy to a Metformin & Saxagliptin Combination in Patients With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ikfe-CRO GmbH (Industry)
Collaborators: AstraZeneca (Industry); IKFE Institute for Clinical Research and Development (Other)
Responsible Party: Prof. Andreas Pfuetzner, IKFE Institute for Clinical Research and Development
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AZ-SAX-001
Record Dates: First submitted 2010-09-15; First posted 2010-09-22 (Estimated); Last update posted 2010-09-22 (Estimated); Status verified 2010-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; saxagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control arm (No Intervention): The patients randomized to the control arm will continue their current therapy, as individually prescribed. Insulin will be administered via subcutaneous injection and OADs (if applicable) will be administered orally, as individually prescribed.
- Saxagliptin & metformin (Experimental): Saxagliptin and metformin tablets will be administered orally. Pioglitazione (Rescue medication) tablets will be administered orally. Insulin glargine (Rescue medication) will be administered via subcutaneous injection as individually prescribed.
  Interventions: Drug: Metformin and Saxagliptin

INTERVENTIONS:
Drug: Metformin and Saxagliptin — Metformin 500mg/daily titrated to 2000mg/d in 4 Weeks (continued for 20 weeks) Saxagliptin 5 mg daily over complete trial
  Arms: Saxagliptin & metformin

SUMMARY:
The purpose of this study is to investigate the success rate of a switch from insulin therapy to a metformin & saxagliptin combination in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
The following study is based on a previous clinical trial performed at ikfe GmbH in Mainz in 2006 and 2007 (PIOswitch). [2] The purpose of this trial was to demonstrate that type 2 diabetes patients treated with insulin can be effectively switched to a pioglitazone/glimepiride combination without loss of glycemic control. The study was performed with 100 patients, out of whom 76 were finally successfully switched, resulting in a cheaper and more convenient therapy with indications of an improved laboratory cardiovascular risk biomarker profile (Hohberg et al., Diabetes Obes. Metab. 11:464-471, 2009). [2] Glimeperide is an agent with unspecific stimulating effect on the ß-cell and is considered to accelerate the progression of the disease while still controlling blood glucose. In addition, it may cause hypoglycemia. The combination of pioglitazone with glimepiride was selected, because pioglitazone requires approx. 5-6 weeks for developing its full anti-diabetic efficacy and an immediate effect on glucose was required to avoid glycemic deterioration.

It is tempting to speculate that the combination of a drug providing ß-cell protection (like saxagliptin) with a drug effectively and rapidly lowering blood glucose through a different mechanism of action (metformin) instead of unspecific ß-cell stimulation would result in an even improved outcome without risk of hypoglycemia. The purpose of this study is to investigate the success rate of a switch from insulin therapy to a metformin & saxagliptin combination in patients with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Combination of OAD and basal insulin treatment (BOT) or intensified conventional therapy (ICT; > 2 injections of basal and prandial) or conventional insulin therapy (CIT; 1 or 2 injections of basal or biphasic)
* HbA1c < 7.5 %
* Age: 18-80 years inclusively
* Duration of insulin therapy > 1 year
* Insulin dose < 120 IU/day
* Fasting C-peptide > 0.6 ng/l
* Fasting glucose ≤ 210 mg/dl
* Full legal, mental and physical ability to give informed consent
* Patient consent that the general physician will be informed of trail participation
* Experience in self measurement of blood glucose > 1 year

Exclusion Criteria:

* Type 1 Diabetes mellitus
* History of drug or alcohol abuse within the last five years prior to screening
* History of severe or multiple allergies
* Progressive fatal disease
* History of significant cardiovascular, respiratory, gastrointestinal, hepatic (ALAT and/or ASAT > 3 times the normal reference range), neurological, psychiatric and/or haematological disease as judged by the investigator
* Renal insufficiency or history of significant renal diseases (creatinine clearance lower than 60 ml/min determined using the Cockroft-Goult equation).
* Contra-indications for study drugs including contraindications for the rescue drugs
* Anamnestic history of hypersensitivity to the study drugs or to drugs with similar chemical structures
* Pregnancy or breast feeding
* Sexually active women of childbearing potential not consistently and correctly practicing birth control by implants, injectables, combined oral contraceptives, hormonal intrauterine devices (IUDs), sexual abstinence or vasectomised partner
* Treatment with any other investigational drug within 3 months prior to screening
* Lack of compliance or other similar reason, that according to investigator, precludes satisfactory participation in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
percentage of patients with stable HbA1c | 26 ± 2 weeks (baseline to postbaseline values) at 4 week intervals

SECONDARY OUTCOMES:
impact of the switch on: | 26 ± 2 weeks (baseline to postbaseline values)
  - Biomarkers of insulin resistance and ß-cell function
impact of the switch on: | 26 ± 2 weeks (baseline to postbaseline values)
  - Biomarkers of cardiovaskular risk
impact of the switch on: | 26 ± 2 weeks (baseline to postbaseline values)
  - Patient treatment satifaction
impact of the switch on: | 26 ± 2 weeks (baseline to postbaseline values)
  - Treatment costs
impact of the switch on: | 26 ± 2 weeks (baseline to postbaseline values)
  - Requirement of 3rd line OAD pioglitazone as rescue drug
impact of the switch on: | 26 ± 2 weeks (baseline to postbaseline values)
  - oral Glucose Tolerance Test (oGTT)
impact of the switch on: | 26 ± 2 weeks (baseline to postbaseline values)
  - Macrophagen activation (in a subpopulation at site 01 ikfe GmbH)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Pfützner, Prof.Dr.Dr., Principal Investigator — IKFE Institute for Clinical Research and Development
Locations (7):
- Germany (7):
  - Diabetologische Schwerpunktpraxis Dr. Lorra / Dr. Bonnermann, Bochum
  - Zentrum für klinische Studien Dresden, GWT-TUD GmbH, Dresden
  - Gemeinschaftspraxis Partner der Gesundheit, Essen
  - IKFE Institute for Clinical Research and Development, Mainz
  - Zentrum für Diabetes und Gefäßerkrankungen, Münster
  - Diabetes Zentrum Neuwied, Neuwied
  - ikfe Studiencenter Potsdam GmbH, Potsdam